CLINICAL TRIAL: NCT05924048
Title: Effect of Reducing the Oxygen Concentration From 5% to 2% on Intracytoplasmic Sperm Injection (ICSI) Outcome
Brief Title: Effect of Reducing the Oxygen Concentration From 5% to 2% on ICSI Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Islamic Center for Population Studies and Research (Other)
Responsible Party: Principal Investigator, Ahmed EL-Sayed Sabry Metwally, Principal Investigator, International Islamic Center for Population Studies and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: O2 level in human embryo
Record Dates: First submitted 2023-06-18; First posted 2023-06-29 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: IVF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of 2% oxygen concentration. (Experimental): Incubate human embryo at 2% oxygen concentration.
  Interventions: Other: Reducing the Oxygen Concentration From 5% to 2%
- Group of 5% oxygen concentration. (No Intervention): Incubate human embryo at 5% oxygen concentration.

INTERVENTIONS:
Other: Reducing the Oxygen Concentration From 5% to 2% — Effect of Reducing the Oxygen Concentration From 5% to 2% in arm 1.
  Arms: Group of 2% oxygen concentration.

SUMMARY:
To assess the effect of reducing the oxygen concentration from 5% to 2% on Intracytoplasmic sperm injection (ICSI) outcome.

DETAILED DESCRIPTION:
Oxygen level plays a critical role in reducing the high level of detrimental reactive oxygen species within cells, influences embryonic gene expression, helps with embryo metabolism of glucose, and enhances embryo development from 2PN to the blastocyst stage, the oxygen concentration in the incubator is an important determinant of the in vitro environment that an embryo encounters. The preimplantation embryo consumes oxygen at a relatively constant level from the one-cell through the morula stage, while at the blastocyst stage the consumption is considerably increased. Oxygen plays a role in energy production, but in too high concentrations it may have a toxic effect by the formation of reactive oxygen species. While in vivo oxygen levels range from 1.5 to 8.7% in the fallopian tubes and uterus of several species, in most laboratories in vitro culture of human embryos was traditionally performed under atmospheric oxygen concentrations (~20%) . In mammals, the oxygen (O2) tension in the uterus is lower (2%) than the oviduct (5-7%). This fits with a shift in the metabolic strategy of the embryo after compaction and may have implications for EC in clinical IVF. Indeed, in a recent study utilizing discarded human embryos, blastulation rates were superior when cultured in 2% compared to 5% after day day 3. However, it is exceedingly difficult to control for the myriad factors impacting blastulation when employing discarded material . The technologies available in the early days of IVF, and most likely also for financial reasons, led to the widespread implementation of incubators that used atmospheric air (i.e. 20% oxygen) . Around the turn of the last century, more advanced incubators capable of creating an environment of 5% oxygen, which better resembles the natural

environment for oocytes and embryos, were developed. Currently, in around 60% of the IVF cycles performed worldwide, the embryos are cultured under 5% oxygen . Kaser et al. add to the long history of experimental data evaluating different oxygen levels in embryo culture. They evaluated the impact of a sequential oxygen tension system (5% oxygen from day 1 to day 3; 2% oxygen from day 3 to day 5) in extended culture . The effect of oxygen level during embryo culture on pregnancy and live birth rates is less straightforward. Although most studies found an improvement in embryo quality when culturing embryos under 5% oxygen . This discrepancy is partly explained by lack of power due to small sample sizes in some studies. When data are pooled in meta-analyses, the overall effect favours culture under 5% oxygen . Another explanation for the inconsistent results among the studies could be due to the differences in duration of exposure, until cleavage or blastocyst stage. When data in the meta-analyses were stratified for duration of culture, there was no effect of oxygen on pregnancy or live birth rates after 2-3 days of culture. After culture to the blastocyst stage, however, culture under 5% oxygen resulted in improved ongoing pregnancy. In the previous studies reported that culture under 5% O2 results in significantly more human surplus embryos reaching the blastocyst stage, as well as a higher proportion of blastocysts consisting of a normal number of cells.

in the human, indirect evidence exists that a low O2 tension of 5% appears to enhance the blastulation rate of surplus embryos .

A reduction in oxygen tension from atmospheric to more physiologic levels is beneficial for the mammalian blastocyst, in terms of a higher cell number and decreased apoptosis, less DNA fragmentation and less oxidative stress. During this highly metabolically active period of growth of the embryo and differentiation into trophectoderm (TE) and inner cell mass (ICM), this decrease in oxygen may protect against oxidative stress .

ELIGIBILITY:
Inclusion Criteria:

- Female age 20-35 years. Oocytes with normal morphology.

Exclusion Criteria:

* Embryo number less than 5. Male factor.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 196 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-27 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Number and grad of embryos which exposed to oxygen concentration 2% . | 1.3 year
  Evaluate embryo quality at day 5

SECONDARY OUTCOMES:
Clinical pregnancy rate for examined subject. | 1.5 Year
  Compare the two arms in clinical pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- International Islamic Center, Cairo, Egypt

REFERENCES:
- [Result] Bahceci M, Ciray HN, Karagenc L, Ulug U, Bener F. Effect of oxygen concentration during the incubation of embryos of women undergoing ICSI and embryo transfer: a prospective randomized study. Reprod Biomed Online. 2005 Oct;11(4):438-43. doi: 10.1016/s1472-6483(10)61136-4. PMID 16274603
- [Result] Bontekoe S, Mantikou E, van Wely M, Seshadri S, Repping S, Mastenbroek S. Low oxygen concentrations for embryo culture in assisted reproductive technologies. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008950. doi: 10.1002/14651858.CD008950.pub2. PMID 22786519
- [Result] Christianson MS, Zhao Y, Shoham G, Granot I, Safran A, Khafagy A, Leong M, Shoham Z. Embryo catheter loading and embryo culture techniques: results of a worldwide Web-based survey. J Assist Reprod Genet. 2014 Aug;31(8):1029-36. doi: 10.1007/s10815-014-0250-z. Epub 2014 Jun 10. PMID 24913025
- [Result] Gomes Sobrinho DB, Oliveira JB, Petersen CG, Mauri AL, Silva LF, Massaro FC, Baruffi RL, Cavagna M, Franco JG Jr. IVF/ICSI outcomes after culture of human embryos at low oxygen tension: a meta-analysis. Reprod Biol Endocrinol. 2011 Nov 1;9:143. doi: 10.1186/1477-7827-9-143. PMID 22044493
- [Result] Guerin P, El Mouatassim S, Menezo Y. Oxidative stress and protection against reactive oxygen species in the pre-implantation embryo and its surroundings. Hum Reprod Update. 2001 Mar-Apr;7(2):175-89. doi: 10.1093/humupd/7.2.175. PMID 11284661
- [Result] Dumoulin JC, Meijers CJ, Bras M, Coonen E, Geraedts JP, Evers JL. Effect of oxygen concentration on human in-vitro fertilization and embryo culture. Hum Reprod. 1999 Feb;14(2):465-9. doi: 10.1093/humrep/14.2.465. PMID 10099995
- [Result] Kaser DJ, Bogale B, Sarda V, Farland LV, Williams PL, Racowsky C. Randomized controlled trial of low (5%) versus ultralow (2%) oxygen for extended culture using bipronucleate and tripronucleate human preimplantation embryos. Fertil Steril. 2018 Jun;109(6):1030-1037.e2. doi: 10.1016/j.fertnstert.2018.02.119. PMID 29935641
- [Result] Kea B, Gebhardt J, Watt J, Westphal LM, Lathi RB, Milki AA, Behr B. Effect of reduced oxygen concentrations on the outcome of in vitro fertilization. Fertil Steril. 2007 Jan;87(1):213-6. doi: 10.1016/j.fertnstert.2006.05.066. Epub 2006 Nov 1. PMID 17081523
- [Result] Kovacic B, Sajko MC, Vlaisavljevic V. A prospective, randomized trial on the effect of atmospheric versus reduced oxygen concentration on the outcome of intracytoplasmic sperm injection cycles. Fertil Steril. 2010 Jul;94(2):511-9. doi: 10.1016/j.fertnstert.2009.03.077. Epub 2009 May 5. PMID 19409544
- [Result] Meintjes M, Chantilis SJ, Douglas JD, Rodriguez AJ, Guerami AR, Bookout DM, Barnett BD, Madden JD. A controlled randomized trial evaluating the effect of lowered incubator oxygen tension on live births in a predominantly blastocyst transfer program. Hum Reprod. 2009 Feb;24(2):300-7. doi: 10.1093/humrep/den368. Epub 2008 Oct 16. PMID 18927130
- [Result] Nastri CO, Nobrega BN, Teixeira DM, Amorim J, Diniz LMM, Barbosa MWP, Giorgi VSI, Pileggi VN, Martins WP. Low versus atmospheric oxygen tension for embryo culture in assisted reproduction: a systematic review and meta-analysis. Fertil Steril. 2016 Jul;106(1):95-104.e17. doi: 10.1016/j.fertnstert.2016.02.037. Epub 2016 Mar 21. PMID 27012651